CLINICAL TRIAL: NCT01961830
Title: An Open-label, Single Dose Study to Assess Intrapulmonary Pharmacokinetics of ME1100 Inhalation Solution Administered to Healthy Volunteers
Brief Title: Intrapulmonary Pharmacokinetics of ME1100 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME1100-CL-102
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — arbekacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ME1100 (Experimental): ME1100 inhalation solution 0.6 mL for 90 mg, Single Dose ME1100 inhalation solution 3.0 mL for 450 mg, Single Dose
  Interventions: Drug: ME1100 inhalation solution

INTERVENTIONS:
Drug: ME1100 inhalation solution
  Other Names: arbekacin

SUMMARY:
This is a single-center, open-label, single-dose study. The primary objective is to determine Epithelial Lining Fluid (ELF) levels of ME1100 after a single orally inhaled dose. The secondary objectives are to determine systemic exposure to inhaled ME1100 and to assess tolerability and safety of a single dose of ME1100 inhalation solution.

ELIGIBILITY:
Inclusion Criteria:

* Male (who are surgically sterile or agree to practice barrier contraception throughout their participation in the study) or Female (using oral, hormonal, or double barrier contraceptive if sexually active, surgically sterile or post-menopausal confirmed by Follicle stimulating hormone(FSH) test)
* Willing to give written informed consent
* 18 to 55 years of age at time of consent Body Mass Index (BMI) of 18-30 kg/m2
* Non-smoker (for at least 6 months prior to screening) and willing to abstain from smoking during the course of the study
* Good general health as determined by medical history, physical examination, Electrocardiogram(ECG) and clinical laboratory tests (including normal renal function and high frequency audiometry)
* Willing to abstain from alcohol, caffeine, and xanthine-containing beverages for 24 hours prior to and 72 hours after dosing.

Exclusion Criteria:

* Uncontrolled, clinically significant disease which in the opinion of the Principal Investigator or Medical Monitor would place the subject at risk through study participation or would confound the assessment of the safety of ME1100 inhalation solution
* Evidence of current or history of respiratory disease, including asthma, emphysema, chronic bronchitis, or cystic fibrosis
* History or current symptom(s) of respiratory tract inflammation within 30 days of Visit 2
* History of hearing, balance or ear disorder or surgery or injury to the ears, or with genetic mutation (>5.0% heteroplasmy) suggestive of increased risk of hearing loss (MT-RNR1 [A1555G] for mitochondrial 12S ribosomal RNA gene or MT-TS1 [A3243G] for mitochondrial transfer RNA serine 1)
* History of parent, sibling or parental sibling reporting hearing loss before age 65 years
* History of malignancy
* History of clinically significant alcohol or drug abuse
* History within last 6 months or current use of any tobacco products including e-cigarettes.
* Positive drug screen for drugs of abuse
* Positive test for HIV, Hepatitis B or Hepatitis C
* Use of any prescription or over-the-counter medications (except oral or hormonal contraceptives), herbal supplements, or vitamins within 14 days of Visit 2
* Known hypersensitivity to any aminoglycoside or lidocaine
* Female of childbearing potential with a positive urine pregnancy test, or currently breast feeding.
* Inability to perform reproducible spirometry in accordance with American Thoracic Society (ATS) guidelines
* Abnormal Forced Expiratory Volume in the First Second(FEV1), Forced Vital Capacity(FVC), or FEV1/FVC (FEV1 or FVC < 80% of predicted or FEV1/FVC ratio < 0.7)
* FEV1 variability > 10% between V1 and V2 (prior to dosing)
* Significant blood donation (or testing) in previous 8 weeks before screening.
* Use of any Investigational Product in previous 30 days or 5 half-lives, whichever is longer, preceding start of screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics profile in ELF | 0-12 hours after START of Dosing
  Each subject will undergo fiber-optic bronchoscopy for the collection of bronchoalveolar lavage fluid at one of the following time points:5 minutes after END of dosing, 0.5, 1, 3, 6 and 12 hrs post START of dosing.

SECONDARY OUTCOMES:
Serum Concentration of ME1100 | 2, 5, 10 minutes after END of dosing, 0.5, 1, 3, 6 and 12 hrs post START of dosing
Number of participants with abnormal safety laboratory measurements | from Baseline to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuharu Egawa, Study Chair — Meiji Seika Pharma Co., Ltd.
Locations (1):
- Pulmonary Associates, Phoenix, Arizona, United States